CLINICAL TRIAL: NCT07019519
Title: Interplay Between Gut Hormones and Autonomic Postprandial Blood Flow Regulation in Patients With POTS
Brief Title: POTS-FLOW: Interplay Between Gut Hormones and Autonomic Postprandial Blood Flow Regulation in Patients With POTS
Acronym: GA22
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H-24030176
Record Dates: First submitted 2025-03-13; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Postural Orthostatic Tachycardia Syndrome (POTS); Healthy
Keywords: Postural Orthostatic Tachycardia Syndrome; POTS; Glucose-dependent insulinotropic polypeptide; GIP; Glucagon-like peptide-1; Glucagon-like peptide-2; GLP-1; GLP-2; CCK-8; Cholecystokinin; Splanchnic Blood Flow
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Single blinded, randomized, crossover trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Saline (Active Comparator): Saline infusion, oral glucose (POTS and healthy)
  Interventions: Other: Saline/Placebo
- GIP antagonist (Experimental): GIP(3-30)NH2 infusion, oral glucose (POTS and healthy)
  Interventions: Other: GIPR antagonist
- GLP-1 antagonist (Experimental): Exendin(9-39)NH2 infusion, oral glucose (only in healthy)
  Interventions: Other: GLP-1R antagonist
- CCK agonist (Experimental): CCK-8 infusion, oral glucose (POTS and healthy)
  Interventions: Other: CCK agonist

INTERVENTIONS:
Other: Saline/Placebo — NaCl(9mg/ml)
  Arms: Saline
Other: GIPR antagonist — GIP(3-30)NH2
  Arms: GIP antagonist
Other: GLP-1R antagonist — GLP-1(9-39)NH2
  Arms: GLP-1 antagonist
Other: CCK agonist — CCK-8
  Arms: CCK agonist

SUMMARY:
This study will describe the interplay between the gut hormones GIP and CCK and their regulation of blood flow to the large vessels in patients with Postural Orthostatic Tachycardia Syndrome (POTS) and GIP, CCK and GLP-1 in healthy. This is addressed by hormone infusions during MR-scans of the abdomen and intake of oral glucose.

DETAILED DESCRIPTION:
Each participant will attend independent randomized experimental days with MR-scans during and intravenous infusions of hormones or placebo and ingestion of glucose or water. A continuous intravenous infusion of either GIP(3-30)NH2, CCK8- or saline for POTS-group or GIP(3-30)NH2, CCK-8, saline or exendin(9-39)NH2 in healthy is started while the participant lie in the scanner while scans, blood samples and questionnaires are repeated over the time course of 2 hours. At a specific timepoint the participants will ingest 75 g of glucose dissolved in 250 ml water.

ELIGIBILITY:
Inclusion Criteria POTS patients:

* Previously diagnosed with POTS in tilt test or active stand-test (either newly diagnosed within last 3 months or in new tilt test/active stand test during screenings visit)
* Reproducible orthostatic intolerance with raise in HR on >30 bpm when standing within 10 minutes of change of supine to standing in age >19 years or >40 bpm in age 18-19 years.
* POTS symptoms/orthostatic intolerance
* Age 18-50
* Waist ratio <180 cm

Exclusion Criteria:

* Chronic illness
* Metallic implants
* Above 10 alcoholic drinks or week or substance abuse
* Other types of sinus tachycardia or heart disease
* Liverenzymes two times above normal values
* Decreased kidney function eGFR <90 or elevated kreatinkinasis
* Thyroid disease or TSH out of reference
* Uncontrollable low or high blood pressure
* Blood vessels that cannot be visualized on MR
* Any disease that might influence the health of the participant during the study or participants that receives medicine that cannot be paused for 36 hours

Inclusion Criteria:

* Age 18-50
* Waist ratio <180 cm
* Matched a POTS patient in age, sex and BMI

Exclusion Criteria:

* Chronic illness
* Metallic implants
* Above 10 alcoholic drinks or week or substance abuse
* POTS; other types of sinus tachycardia or heart disease
* Liverenzymes two times above normal values
* Decreased kidney function eGFR <90 or elevated kreatinkinasis
* Thyroid disease or TSH out of reference
* Uncontrollable low or high blood pressure, Orthostatic hypotension
* Blood vessels that cannot be visualized on MR
* Any disease that might influence the health of the participant during the study or participants that receives medicine that cannot be paused for 36 hours

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Redistribution of splanchnic blood flow in the vessel mesenteric superior artery (MR) | Continuously for 80 minutes/during infusions
  Blood flow in the superior mesenteric artery measured with MR ml/min

SECONDARY OUTCOMES:
Blood flow in portal vein | Continuously for 80 minutes/during infusions
  Blood flow in the portal vein measured with MR-scans in ml/min
Blood Flow in celiac trunk | Continuously for 80 minutes/during infusions
  Blood flow in the celiac trunk measured with MR-scans in ml/min
Blood Flow in the hepatic artery | Continuously for 80 minutes/during infusions
  Blood flow in the hepatic artery measured with MR-scans in ml/min
Blood samples for hormones | Every 10-20 minutes before and during and after the infusions and MR scans (120 minutes)
  Blood samples of hormones types:
  GLP-1(7-36 NH2), GLP-2(1-33), GIP(1-42), Exendin(9-39)NH2, GLP-2(3-33), GIP(3-30)NH2, Glucagon, Insulin/C-peptid, CCK
Gastric emptying/Blood sample of paracetamol | Every 10-20 minutes before, during and after the infusions and MRI scans (120 minutes)
  Uptake/amount of paracetamol in the blood over time as a measure of gastric emptying
Symptomscoring | Continously before and during the infusions (120 minutes)
  Symptomscoring of autonome dysfunction with VOSS (Vanderbilt Orthostatic Symptom Score) questionnaire: this consists of 10 symptoms: lightheadedness, brain fog, shortness of breath, palpitations, tremor, headache, tightness in chest, blurred vision, nausea and sleepiness rated from 0-10 where 0 is not ocurring and 10 is worts experienced.
Blood samples for genes | One measurement at baseline visit
  Genes analyzed from buffycoat:
  GLP-1R: NM_002062, GLP-2R: NM_004246, GIPR: NM_000164 and NM_001308418, CCKR: NM_000730 and NM_176875,
Blood sample for glucose | Every 10-20 minutes before and during and after the infusions and MR scans (120 minutes)
  Glucose measurements
Blood samples for autoantibodies | One measurement at baseline visit
  Autoantibodies:
  Angiotensin-II-receptor-1 AT1R-ab, Endothelin-receptor-A ETAR-ab, Alpha1 adrenergic-receptor-ab, Alpha2 adrenergic-receptor-ab, Beta1 adrenergic-receptor-ab, Beta2 adrenergic-receptor-ab, Muscarinic cholinergic M1-receptor-ab, Muscarinic cholinergic M2-receptor-ab, Muscarinic cholinergic M3-receptor-ab, Muscarinic cholinergic M4-receptor-ab, Muscarinic cholinergic M5-receptor-ab

CONTACTS AND LOCATIONS:
Overall Officials: Lærke S Gasbjerg, MD, PhD, Study Chair — University of Copenhagen, Rigshospitalet
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Will share upon request
Supporting Information: SAP
Time Frame: Data will be shared upon request after study completion
Access Criteria: Qualified researchers can request access by submitting a proposal to the study sponsor. Data will be shared via a secure online repository upon approval of the request.

REFERENCES:
- [Background] Someya N, Endo MY, Fukuba Y, Hayashi N. Blood flow responses in celiac and superior mesenteric arteries in the initial phase of digestion. Am J Physiol Regul Integr Comp Physiol. 2008 Jun;294(6):R1790-6. doi: 10.1152/ajpregu.00553.2007. Epub 2008 Apr 2. PMID 18385466
- [Background] Parker DR, Carlisle K, Cowan FJ, Corrall RJ, Read AE. Postprandial mesenteric blood flow in humans: relationship to endogenous gastrointestinal hormone secretion and energy content of food. Eur J Gastroenterol Hepatol. 1995 May;7(5):435-40. PMID 7614106
- [Background] Randall EB, Billeschou A, Brinth LS, Mehlsen J, Olufsen MS. A model-based analysis of autonomic nervous function in response to the Valsalva maneuver. J Appl Physiol (1985). 2019 Nov 1;127(5):1386-1402. doi: 10.1152/japplphysiol.00015.2019. Epub 2019 Aug 1. PMID 31369335
- [Background] Mehr SE, Barbul A, Shibao CA. Gastrointestinal symptoms in postural tachycardia syndrome: a systematic review. Clin Auton Res. 2018 Aug;28(4):411-421. doi: 10.1007/s10286-018-0519-x. Epub 2018 Mar 16. PMID 29549458
- [Background] Breier NC, Paranjape SY, Scudder S, Mehr SE, Diedrich A, Flynn CR, Okamoto LE, Hartmann B, Gasbjerg LS, Shibao CA. Worsening Postural Tachycardia Syndrome Is Associated With Increased Glucose-Dependent Insulinotropic Polypeptide Secretion. Hypertension. 2022 May;79(5):e89-e99. doi: 10.1161/HYPERTENSIONAHA.121.17852. Epub 2022 Mar 2. PMID 35232225
- [Background] Koffert J, Honka H, Teuho J, Kauhanen S, Hurme S, Parkkola R, Oikonen V, Mari A, Lindqvist A, Wierup N, Groop L, Nuutila P. Effects of meal and incretins in the regulation of splanchnic blood flow. Endocr Connect. 2017 Apr;6(3):179-187. doi: 10.1530/EC-17-0015. Epub 2017 Mar 3. PMID 28258126
- [Background] Asmar M, Asmar A, Simonsen L, Gasbjerg LS, Sparre-Ulrich AH, Rosenkilde MM, Hartmann B, Dela F, Holst JJ, Bulow J. The Gluco- and Liporegulatory and Vasodilatory Effects of Glucose-Dependent Insulinotropic Polypeptide (GIP) Are Abolished by an Antagonist of the Human GIP Receptor. Diabetes. 2017 Sep;66(9):2363-2371. doi: 10.2337/db17-0480. Epub 2017 Jun 30. PMID 28667118
- [Background] Asmar M, Simonsen L, Madsbad S, Stallknecht B, Holst JJ, Bulow J. Glucose-dependent insulinotropic polypeptide may enhance fatty acid re-esterification in subcutaneous abdominal adipose tissue in lean humans. Diabetes. 2010 Sep;59(9):2160-3. doi: 10.2337/db10-0098. Epub 2010 Jun 14. PMID 20547981
- [Background] Zadourian A, Doherty TA, Swiatkiewicz I, Taub PR. Postural Orthostatic Tachycardia Syndrome: Prevalence, Pathophysiology, and Management. Drugs. 2018 Jul;78(10):983-994. doi: 10.1007/s40265-018-0931-5. PMID 29943373
- [Background] Shaw BH, Stiles LE, Bourne K, Green EA, Shibao CA, Okamoto LE, Garland EM, Gamboa A, Diedrich A, Raj V, Sheldon RS, Biaggioni I, Robertson D, Raj SR. The face of postural tachycardia syndrome - insights from a large cross-sectional online community-based survey. J Intern Med. 2019 Oct;286(4):438-448. doi: 10.1111/joim.12895. Epub 2019 Apr 16. PMID 30861229
- [Background] Freeman R, Wieling W, Axelrod FB, Benditt DG, Benarroch E, Biaggioni I, Cheshire WP, Chelimsky T, Cortelli P, Gibbons CH, Goldstein DS, Hainsworth R, Hilz MJ, Jacob G, Kaufmann H, Jordan J, Lipsitz LA, Levine BD, Low PA, Mathias C, Raj SR, Robertson D, Sandroni P, Schatz I, Schondorff R, Stewart JM, van Dijk JG. Consensus statement on the definition of orthostatic hypotension, neurally mediated syncope and the postural tachycardia syndrome. Clin Auton Res. 2011 Apr;21(2):69-72. doi: 10.1007/s10286-011-0119-5. No abstract available. PMID 21431947
- [Background] Thomsen RW, Ozturk B, Pedersen L, Nicolaisen SK, Petersen I, Olsen J, Sorensen HT. Hospital Records of Pain, Fatigue, or Circulatory Symptoms in Girls Exposed to Human Papillomavirus Vaccination: Cohort, Self-Controlled Case Series, and Population Time Trend Studies. Am J Epidemiol. 2020 Apr 2;189(4):277-285. doi: 10.1093/aje/kwz284. PMID 31899791
- [Background] Mar PL, Raj SR. Postural Orthostatic Tachycardia Syndrome: Mechanisms and New Therapies. Annu Rev Med. 2020 Jan 27;71:235-248. doi: 10.1146/annurev-med-041818-011630. Epub 2019 Aug 14. PMID 31412221
- [Background] Stewart JM, Medow MS, Glover JL, Montgomery LD. Persistent splanchnic hyperemia during upright tilt in postural tachycardia syndrome. Am J Physiol Heart Circ Physiol. 2006 Feb;290(2):H665-73. doi: 10.1152/ajpheart.00784.2005. Epub 2005 Sep 2. PMID 16143646
- [Background] Stewart JM, Montgomery LD. Regional blood volume and peripheral blood flow in postural tachycardia syndrome. Am J Physiol Heart Circ Physiol. 2004 Sep;287(3):H1319-27. doi: 10.1152/ajpheart.00086.2004. Epub 2004 Apr 29. PMID 15117717
- [Background] Stewart JM, Pianosi P, Shaban MA, Terilli C, Svistunova M, Visintainer P, Medow MS. Postural Hyperventilation as a Cause of Postural Tachycardia Syndrome: Increased Systemic Vascular Resistance and Decreased Cardiac Output When Upright in All Postural Tachycardia Syndrome Variants. J Am Heart Assoc. 2018 Jun 30;7(13):e008854. doi: 10.1161/JAHA.118.008854. PMID 29960989
- [Background] Tani H, Singer W, McPhee BR, Opfer-Gehrking TL, Haruma K, Kajiyama G, Low PA. Splanchnic-mesenteric capacitance bed in the postural tachycardia syndrome (POTS). Auton Neurosci. 2000 Dec 28;86(1-2):107-13. doi: 10.1016/S1566-0702(00)00205-8. PMID 11269915
- [Background] Jacob G, Costa F, Shannon JR, Robertson RM, Wathen M, Stein M, Biaggioni I, Ertl A, Black B, Robertson D. The neuropathic postural tachycardia syndrome. N Engl J Med. 2000 Oct 5;343(14):1008-14. doi: 10.1056/NEJM200010053431404. PMID 11018167
- [Background] Mustafa HI, Garland EM, Biaggioni I, Black BK, Dupont WD, Robertson D, Raj SR. Abnormalities of angiotensin regulation in postural tachycardia syndrome. Heart Rhythm. 2011 Mar;8(3):422-8. doi: 10.1016/j.hrthm.2010.11.009. Epub 2011 Jan 22. PMID 21266211
- [Background] Knoop I, Picariello F, Jenkinson E, Gall N, Chisari C, Moss-Morris R. Self-reported symptom burden in postural orthostatic tachycardia syndrome (POTS): A narrative review of observational and interventional studies. Auton Neurosci. 2023 Jan;244:103052. doi: 10.1016/j.autneu.2022.103052. Epub 2022 Nov 18. PMID 36525900
- [Background] Pugliese D, Ohnishi K, Tsunoda T, Sabba C, Albano O. Portal hemodynamics after meal in normal subjects and in patients with chronic liver disease studied by echo-Doppler flowmeter. Am J Gastroenterol. 1987 Oct;82(10):1052-6. PMID 2959148
- [Background] Norryd C, Denker H, Lunderquist A, Olin T, Tylen U. Superior mesenteric blood flow during digestion in man. Acta Chir Scand. 1975;141(3):197-202. PMID 1166743
- [Background] Takala J. Determinants of splanchnic blood flow. Br J Anaesth. 1996 Jul;77(1):50-8. doi: 10.1093/bja/77.1.50. No abstract available. PMID 8703630
- [Background] Parsonage W, Hetmanski D, Cowley A. Differentiation of the metabolic and vascular effects of insulin in insulin resistance in patients with chronic heart failure. Am J Cardiol. 2002 Mar 15;89(6):696-703. doi: 10.1016/s0002-9149(01)02342-6. PMID 11897212
- [Background] Bremholm L, Andersen UB, Hornum M, Hilsted L, Veedfald S, Hartmann B, Holst JJ. Acute effects of glucagon-like peptide-1, GLP-19-36 amide, and exenatide on mesenteric blood flow, cardiovascular parameters, and biomarkers in healthy volunteers. Physiol Rep. 2017 Feb;5(4):e13102. doi: 10.14814/phy2.13102. PMID 28235974
- [Background] Waaler BA, Eriksen M. Post-prandial cardiovascular responses in man after ingestion of carbohydrate, protein or fat. Acta Physiol Scand. 1992 Nov;146(3):321-7. doi: 10.1111/j.1748-1716.1992.tb09426.x. PMID 1481689
- [Background] Zreik F, Meshulam R, Shichel I, Webb M, Shibolet O, Jacob G. Effect of ingesting a meal and orthostasis on the regulation of splanchnic and systemic hemodynamics and the responsiveness of cardiovascular alpha1-adrenoceptors. Am J Physiol Gastrointest Liver Physiol. 2021 Nov 1;321(5):G513-G526. doi: 10.1152/ajpgi.00142.2021. Epub 2021 Sep 15. PMID 34523347
- [Background] Haddock BT, Francis ST, Larsson HBW, Andersen UB. Assessment of Perfusion and Oxygenation of the Human Renal Cortex and Medulla by Quantitative MRI during Handgrip Exercise. J Am Soc Nephrol. 2018 Oct;29(10):2510-2517. doi: 10.1681/ASN.2018030272. Epub 2018 Sep 11. PMID 30206141
- [Background] Haddock B, Larsson HBW, Francis S, Andersen UB. Human renal response to furosemide: Simultaneous oxygenation and perfusion measurements in cortex and medulla. Acta Physiol (Oxf). 2019 Sep;227(1):e13292. doi: 10.1111/apha.13292. Epub 2019 May 21. PMID 31046189
- [Background] Ban K, Noyan-Ashraf MH, Hoefer J, Bolz SS, Drucker DJ, Husain M. Cardioprotective and vasodilatory actions of glucagon-like peptide 1 receptor are mediated through both glucagon-like peptide 1 receptor-dependent and -independent pathways. Circulation. 2008 May 6;117(18):2340-50. doi: 10.1161/CIRCULATIONAHA.107.739938. Epub 2008 Apr 21. PMID 18427132
- [Background] Xiong QF, Fan SH, Li XW, Niu Y, Wang J, Zhang X, Chen YF, Shi YW, Zhang LH. GLP-1 Relaxes Rat Coronary Arteries by Enhancing ATP-Sensitive Potassium Channel Currents. Cardiol Res Pract. 2019 Oct 23;2019:1968785. doi: 10.1155/2019/1968785. eCollection 2019. PMID 31772770
- [Background] Asmar A, Asmar M, Simonsen L, Madsbad S, Holst JJ, Hartmann B, Sorensen CM, Bulow J. Glucagon-like peptide-1 elicits vasodilation in adipose tissue and skeletal muscle in healthy men. Physiol Rep. 2017 Feb;5(3):e13073. doi: 10.14814/phy2.13073. PMID 28174344
- [Background] Bremholm L, Hornum M, Henriksen BM, Larsen S, Holst JJ. Glucagon-like peptide-2 increases mesenteric blood flow in humans. Scand J Gastroenterol. 2009;44(3):314-9. doi: 10.1080/00365520802538195. PMID 19005872
- [Background] Yusta B, Matthews D, Flock GB, Ussher JR, Lavoie B, Mawe GM, Drucker DJ. Glucagon-like peptide-2 promotes gallbladder refilling via a TGR5-independent, GLP-2R-dependent pathway. Mol Metab. 2017 Mar 31;6(6):503-511. doi: 10.1016/j.molmet.2017.03.006. eCollection 2017 Jun. PMID 28580281
- [Background] Drucker DJ, Yusta B. Physiology and pharmacology of the enteroendocrine hormone glucagon-like peptide-2. Annu Rev Physiol. 2014;76:561-83. doi: 10.1146/annurev-physiol-021113-170317. Epub 2013 Oct 25. PMID 24161075
- [Background] Kogire M, Inoue K, Sumi S, Doi R, Takaori K, Yun M, Fujii N, Yajima H, Tobe T. Effects of synthetic human gastric inhibitory polypeptide on splanchnic circulation in dogs. Gastroenterology. 1988 Dec;95(6):1636-40. doi: 10.1016/s0016-5085(88)80089-1. PMID 3053315
- [Background] Sartor DM, Verberne AJ. Abdominal vagal signalling: a novel role for cholecystokinin in circulatory control? Brain Res Rev. 2008 Nov;59(1):140-54. doi: 10.1016/j.brainresrev.2008.07.002. Epub 2008 Jul 12. PMID 18656498
- [Background] Sieber C, Beglinger C, Jaeger K, Hildebrand P, Stalder GA. Regulation of postprandial mesenteric blood flow in humans: evidence for a cholinergic nervous reflex. Gut. 1991 Apr;32(4):361-6. doi: 10.1136/gut.32.4.361. PMID 2026334
- [Background] Gilliam-Vigh H, Jorsal T, Rehfeld JF, Pedersen J, Poulsen SS, Vilsboll T, Knop FK. Expression of Cholecystokinin and its Receptors in the Intestinal Tract of Type 2 Diabetes Patients and Healthy Controls. J Clin Endocrinol Metab. 2021 Jul 13;106(8):2164-2170. doi: 10.1210/clinem/dgab367. PMID 34036343
- [Background] Lynggaard MB, Gasbjerg LS, Christensen MB, Knop FK. GIP(3-30)NH2 - a tool for the study of GIP physiology. Curr Opin Pharmacol. 2020 Dec;55:31-40. doi: 10.1016/j.coph.2020.08.011. Epub 2020 Oct 11. PMID 33053504
- [Background] Melchiorsen JU, Sorensen KV, Bork-Jensen J, Kizilkaya HS, Gasbjerg LS, Hauser AS, Rungby J, Sorensen HT, Vaag A, Nielsen JS, Pedersen O, Linneberg A, Hartmann B, Gjesing AP, Holst JJ, Hansen T, Rosenkilde MM, Grarup N. Rare Heterozygous Loss-of-Function Variants in the Human GLP-1 Receptor Are Not Associated With Cardiometabolic Phenotypes. J Clin Endocrinol Metab. 2023 Oct 18;108(11):2821-2833. doi: 10.1210/clinem/dgad290. PMID 37235780
- [Background] Buttner J, Bluthner E, Greif S, Kuhl A, Elezkurtaj S, Ulrich J, Maasberg S, Jochum C, Tacke F, Pape UF. Predictive Potential of Biomarkers of Intestinal Barrier Function for Therapeutic Management with Teduglutide in Patients with Short Bowel Syndrome. Nutrients. 2023 Sep 29;15(19):4220. doi: 10.3390/nu15194220. PMID 37836505
- [Background] Wank SA, Pisegna JR, de Weerth A. Cholecystokinin receptor family. Molecular cloning, structure, and functional expression in rat, guinea pig, and human. Ann N Y Acad Sci. 1994 Mar 23;713:49-66. doi: 10.1111/j.1749-6632.1994.tb44052.x. PMID 8185215
- [Background] Cox EF, Palaniyappan N, Aithal GP, Guha IN, Francis ST. Using MRI to study the alterations in liver blood flow, perfusion, and oxygenation in response to physiological stress challenges: Meal, hyperoxia, and hypercapnia. J Magn Reson Imaging. 2019 Jun;49(6):1577-1586. doi: 10.1002/jmri.26341. Epub 2018 Oct 24. PMID 30353969
- [Background] Medhus AW, Lofthus CM, Bredesen J, Husebye E. Gastric emptying: the validity of the paracetamol absorption test adjusted for individual pharmacokinetics. Neurogastroenterol Motil. 2001 Jun;13(3):179-85. doi: 10.1046/j.1365-2982.2001.00249.x. PMID 11437980
- [Background] Deacon CF. Circulation and degradation of GIP and GLP-1. Horm Metab Res. 2004 Nov-Dec;36(11-12):761-5. doi: 10.1055/s-2004-826160. PMID 15655705
- [Background] Deacon CF, Nauck MA, Meier J, Hucking K, Holst JJ. Degradation of endogenous and exogenous gastric inhibitory polypeptide in healthy and in type 2 diabetic subjects as revealed using a new assay for the intact peptide. J Clin Endocrinol Metab. 2000 Oct;85(10):3575-81. doi: 10.1210/jcem.85.10.6855. PMID 11061504
- [Background] Hartmann B, Harr MB, Jeppesen PB, Wojdemann M, Deacon CF, Mortensen PB, Holst JJ. In vivo and in vitro degradation of glucagon-like peptide-2 in humans. J Clin Endocrinol Metab. 2000 Aug;85(8):2884-8. doi: 10.1210/jcem.85.8.6717. PMID 10946898
- [Background] Yamazaki K, Kagaya T, Watanabe M, Terauchi H, Iida D, Fukumoto H, Suzuki S, Arai T, Aoki M, Takase K, Seiki T, Tsukahara K, Nagakawa J. A novel truncated glucagon-like peptide 2 (GLP-2) as a tool for analyzing GLP-2 receptor agonists. Biomed Res. 2013 Jun;34(3):129-36. doi: 10.2220/biomedres.34.129. PMID 23782746
- [Background] Thulesen J, Knudsen LB, Hartmann B, Hastrup S, Kissow H, Jeppesen PB, Orskov C, Holst JJ, Poulsen SS. The truncated metabolite GLP-2 (3-33) interacts with the GLP-2 receptor as a partial agonist. Regul Pept. 2002 Jan 15;103(1):9-15. doi: 10.1016/s0167-0115(01)00316-0. PMID 11738243
- [Background] Hansen LS, Sparre-Ulrich AH, Christensen M, Knop FK, Hartmann B, Holst JJ, Rosenkilde MM. N-terminally and C-terminally truncated forms of glucose-dependent insulinotropic polypeptide are high-affinity competitive antagonists of the human GIP receptor. Br J Pharmacol. 2016 Mar;173(5):826-38. doi: 10.1111/bph.13384. Epub 2016 Jan 30. PMID 26572091
- [Background] Gasbjerg LS, Christensen MB, Hartmann B, Lanng AR, Sparre-Ulrich AH, Gabe MBN, Dela F, Vilsboll T, Holst JJ, Rosenkilde MM, Knop FK. GIP(3-30)NH2 is an efficacious GIP receptor antagonist in humans: a randomised, double-blinded, placebo-controlled, crossover study. Diabetologia. 2018 Feb;61(2):413-423. doi: 10.1007/s00125-017-4447-4. Epub 2017 Sep 25. PMID 28948296
- [Background] Schjoldager BT. Role of CCK in gallbladder function. Ann N Y Acad Sci. 1994 Mar 23;713:207-18. doi: 10.1111/j.1749-6632.1994.tb44067.x. PMID 8185161
- [Background] Rohde U, Sonne DP, Christensen M, Hansen M, Bronden A, Torang S, Rehfeld JF, Holst JJ, Vilsboll T, Knop FK. Cholecystokinin-Induced Gallbladder Emptying and Metformin Elicit Additive Glucagon-Like Peptide-1 Responses. J Clin Endocrinol Metab. 2016 May;101(5):2076-83. doi: 10.1210/jc.2016-1133. Epub 2016 Mar 22. PMID 27003305
- [Background] Ruiz-Gayo M, Gonzalez MC, Fernandez-Alfonso S. Vasodilatory effects of cholecystokinin: new role for an old peptide? Regul Pept. 2006 Dec 10;137(3):179-84. doi: 10.1016/j.regpep.2006.06.006. Epub 2006 Aug 2. PMID 16889840
- [Background] Sheldon RS, Grubb BP 2nd, Olshansky B, Shen WK, Calkins H, Brignole M, Raj SR, Krahn AD, Morillo CA, Stewart JM, Sutton R, Sandroni P, Friday KJ, Hachul DT, Cohen MI, Lau DH, Mayuga KA, Moak JP, Sandhu RK, Kanjwal K. 2015 heart rhythm society expert consensus statement on the diagnosis and treatment of postural tachycardia syndrome, inappropriate sinus tachycardia, and vasovagal syncope. Heart Rhythm. 2015 Jun;12(6):e41-63. doi: 10.1016/j.hrthm.2015.03.029. Epub 2015 May 14. No abstract available. PMID 25980576

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT07019519/Prot_SAP_000.pdf